CLINICAL TRIAL: NCT00006214
Title: Short-Term Chemoprevention Trial in Men With Prostatic Intraepithelial Neoplasia Using Flutamide as an Androgen Deprivation Agent
Brief Title: Flutamide In the Prevention of Prostate Cancer in Patients With Neoplasia of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCCTG-959257; CDR0000067929 (Registry Identifier: PDQ (Physician Data Query)); MAYO-959257; MAYO-IRB-921-97; NCI-P00-0156
Record Dates: First submitted 2000-09-11; First posted 2004-06-22 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- flutamide (Experimental): Patients receive oral flutamide once daily.
  Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before study, at 1, 6, and 12 months, and then annually therafter. Patients are followed annually for up to 10 years.
  Interventions: Drug: flutamide
- placebo (Other): Patients receive an oral placebo once daily.
  Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before study, at 1, 6, and 12 months, and then annually therafter. Patients are followed annually for up to 10 years.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: flutamide
  Arms: flutamide
Other: placebo
  Arms: placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs such as flutamide to try to prevent the development of cancer. Flutamide may be effective in the prevention of prostate cancer.

PURPOSE: Randomized clinical trial to study the effectiveness of flutamide in preventing prostate cancer in patients who have neoplasia of the prostate.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the ability of flutamide to reduce the incidence of prostate cancer in patients with high grade prostatic intraepithelial neoplasia. II. Determine the effect of this regimen on a series of endpoint biomarkers in these patients. III. Assess the quality of life of these patients.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to age (under 65 versus 65 and over), PSA (0-2.5 versus 2.6-4.0 versus 4.1-10 versus greater than 10 ng/mL), PIN (on one biopsy versus on two biopsies), and family history (prostate cancer in brother, father, or uncle versus no prostate cancer in these relatives). Patients are randomized to one of two treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed high grade prostatic intraepithelial neoplasia Confirmed by second prostate biopsy within 180 days of first biopsy No prior or concurrent prostatic carcinoma No prior hormonal replacement or antiandrogen therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Greater than 5 years Hematopoietic: Not specified Hepatic: SGOT and alkaline phosphatase no greater than 2 times upper limit of normal No hepatitis B or C or liver cirrhosis Renal: Not specified Other: Fertile patients must use effective contraception No other prior malignancy in past 5 years except carcinoma in situ or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: See Disease Characteristics Radiotherapy: No prior radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2000-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Determine the ability of flutamide to reduce the incidence of prostate cancer | Up to 10 years

SECONDARY OUTCOMES:
Overall survival | Up to 10 years
Assess the quality of life of these patients | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (23):
- United States (22):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada